CLINICAL TRIAL: NCT06613906
Title: Efficacy and Safety of Healsea® Isotonic Nasal Spray in the Prevention of Upper Respiratory Tract Infections With Nasal Symptoms in Adults: a Pre-market Study
Brief Title: Prevention With Healsea in Adults Against Respiratory Infection Study
Acronym: PHARIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lallemand Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LPH-2401; 2833/06/08/2024 (Other: Republic of Bulgaria. Ethics Committee for clinical trials)
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Healthy Subjects (HS)
Keywords: saline nasal spray; upper respiratory tract infection; prevention
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healsea Children treated group (Experimental): Subjects of this arm will be treated with Healsea Children nasal spray during 3 treatment periods of 28 days interspersed by 2 wash-out periods of 10 days
- Untreated arm (No Intervention): Subjects of this arm will not receive any treatment for the prevention of respiratory tract infection.

INTERVENTIONS:
Device: Healsea Children nasal spray — dosage: 1 puff in each nostril twice daily during 3 treatment periods of 28 days interspersed by 2 wash-out periods of 10 days

SUMMARY:
Healsea® Children is a class IIa medical device. This is an isotonic seawater-based nasal spray supplemented with a natural Symbiofilm™ extract (0.02%) isolated from marine bacteria. Healsea® Children is indicated in children above 6 years to clean and moisten the nose during colds.

Symbiofilm™, which is not a medicinal product is able to protect the nasal mucosa from viruses entrance by forming a protective barrier on the nasal mucosa.

By targeting the nose as entry points for viruses, we hypothesise that Healsea® Children used regularly during the respiratory virus season may prevent upper respiratory tracts infections such as cold or flu with nasal symptoms not only in children (HEALSPIC study, NCT06582589) but also in adults.

The main objective of this premarket clinical investigation is thus to assess the efficacy of Healsea® Children to prevent upper respiratory tract infections with nasal symptoms in healthy adults during 3 treatment periods of 28 days interspersed by 2 wash-out periods of 10 days when compared to adults not taking Healsea® Children.

198 adults will be randomised in the study, 99 in the Healsea® Children group and 99 in the non-treated group.

The subjects will be asked to report the upper respiratory tract infections with nasal symptoms and complication they may have during the study to the physician in charge of the study conduct.

Two study visits and 3 telephone calls are scheduled. The subjects will also complete an electronic diary to report nasal symptoms and adverse events other than upper respiratory tracts infections.

DETAILED DESCRIPTION:
Upper respiratory tract infections (URTIs) and sino-nasal symptoms are very frequent.

Human rhinovirus (more than 100 serotypes) is the most common cause, accounting up to 50% viral rhinitis episodes in children and adults. These episodes can last up to 7-10 days and are usually self-limited. Prevalence of acute rhinosinusitis varies with season (higher in the fall and winter months) and climatic variations and increases with a damp environment and air pollution. The incidence of acute rhinitis/rhinosinusitis is very high, estimated to occur from 2 to 5 times per year in the average adult.

Healsea® Children is a class IIa medical device. This is an isotonic seawater-based nasal spray supplemented with a natural Symbiofilm™ extract (0.02%) isolated from marine bacteria. Healsea® Children is indicated in children above 6 years to clean and moisten the nose during colds and rhinitis. The clinical performance of Healsea® Children is supported by the sea water solution and Symbiofilm™. The exact mechanisms by which nasal irrigation works are not known. However, most of the experts agree that it is primarily a mechanical intervention leading to direct cleaning of the nasal mucosa.

The other component of Healsea® Children, Symbiofilm™ is an exopolymeric composition with emulsifying/surfactant properties which enhance the cleansing and moistening of nasal mucosa. Furthermore, a prophylactic activity of Symbiofilm™ against infection by viruses involved in upper respiratory infections i.e., Adenovirus, Rhinovirus, Flu virus and OC 43 Coronavirus has been demonstrated in vitro on human nasal epithelial cells (HNEpC). The antiviral prophylactic activity of Symbiofilm™ is suggested to rely on its physiochemical properties that, by coating the surface of epithelial cells, hinders the viral entry process, thus explaining the reduced viral adsorption and the subsequent reduced onset of infection.

By targeting the nose as entry points for viruses, we hypothesise that Healsea® Children used regularly during the respiratory virus season may prevent upper respiratory tracts infections with nasal symptoms not only in children (HEALSPIC study, NCT06582589) but also in the adult population.

The aim of this two arms prospective randomized open-labelled pre-market clinical investigation, is to establish clinical benefits and clinical safety of Healsea® Children to prevent upper respiratory tract infections with nasal symptoms in healthy adults during 3 treatment periods of 28 days (one puff in each ostril twice daily) interspersed by 2 wash-out periods of 10 days when compared to adults not taking Healsea® Children.

198 children will be randomised in the study, 99 in the Healsea® Children group and 99 in the non-treated group.

The subjects will be asked to immediately call the investigator in case of nasal symptoms and complication of respiratory infection they may have during the study.

Two study visits (Visit 1, Screening/Randomisation at Day 1 and Visit 2, End of study visit at Day 106 up to Day 116) and 3 telephone calls (telephone call 1 TC1 at Day15 ±3 days, TC2 at Day 55 ±3 days and TC3 at Day 95±3days) are scheduled. The subjects will also complete an electronic diary to report nasal symptoms, device deficiencies, and adverse events other than upper respiratory tracts infections from D2 up to end of study (Day 106 up to Day 116).

The duration of patient's participation is up to 116 days.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled if they meet all the following criteria:

1. Healthy Male/Female subjects ≥18 years
2. No respiratory tract infection within 15 days before trial entry and at trial entry
3. Willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the information consent form
4. Availability of a smartphone throughout the study and an internet connection.

Exclusion Criteria:

Subjects will not be enrolled if one of the following criteria is present:

1. Known hypersensitivity/allergy to any component of the test device
2. Subject with COPD, severe asthma, perennial allergy, immunodeficiency or cystic fibrosis
3. Body temperature ≥ 37.8°C
4. Medical history or any current disease that is considered by the investigator as a reason for non-inclusion
5. Severe nasal septum deviation or other condition that could cause nasal obstruction such as the presence of nasal polyps
6. Antibiotic (systemic or per nasal route) or antivirals (systemic) intake within 2 weeks before screening
7. Systemic or local corticosteroids (nasal route or inhalation) within 4 weeks before screening
8. Antihistamines intake for allergy when treatment was started from less than 4 weeks before screening
9. Vaccination against flu or COVID-19 within 6 months before screening
10. Chronic decongestant use within 2 weeks before screening
11. Bacterial lysates, or immunostimulants (food supplements excluded) used for prevention of infection within the 6 months before the screening
12. Prebiotics, probiotics used for prevention of infection within 6 months before the screening
13. Pregnant/Lactating female or of childbearing potential without hormonal contraception or intrauterine device or double barrier method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects without any upper respiratory tract infection (URTI) with nasal symptoms during the study. | From the randomization up to Day 116
  The upper respiratory tracts infections with nasal symptoms (blocked nose, runny nose yellow or green discharge, sneezing ) will be collected for each subject throughout the study. An URTI episode with nasal symptoms is defined as follows: (i) at least 1 of the followings must be present: a blocked nose, runny nose, yellow or green nasal discharge, sneezing; (ii) the symptomatic episode must last for at least 3 days.

SECONDARY OUTCOMES:
Number of Upper Respiratory Tract Infections with nasal symptoms during the study | Time Frame: From the randomization up to Day 116
  Upper Respiratory Tract Infections with nasal symptoms will be reported by the subjects to the investigators during the whole study duration and the total number compared between groups
Number of Upper Respiratory Tract Infections complications | Time Frame: From the randomization up to Day 116
  Complications of Upper respiratory Tract Infections (bronchitis, bronchiolitis, pneumoniae, pharyngo-tonsillitis, laryngitis, acute otitis) will be reported by the subjects during the whole study duration and compared between groups
Number of days of use of concomitant treatments that may affect Upper Respiratory Tract Infections symptoms and associated complications | From the randomization up to Day 116
  The number of days of antipyretics intake, systemic or local mucolytics, decongestants, antitussives, systemic and per nasal route antibiotics, local and systemic corticosteroids, systemic antivirals) will be compared between the 2 arms
Number of school days lost due to Upper Respiratory Tract Infections and complications | From the randomization up to Day 116
  Number of school days lost due to Upper Respiratory Tract Infections and complications will be collected during the whole study duration and compared between groups
Assessment of (serious) adverse events and device deficiences throughout the study | From the randomization up to Day 116

CONTACTS AND LOCATIONS:
Locations (1):
- Diagnostics and Consultation Center Convex EOOD,, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williamson S, Dennison L, Greenwell K, Denison-Day J, Mowbray F, Richards-Hall S, Smith D, Bradbury K, Ainsworth B, Little P, Geraghty AWA, Yardley L. Using nasal sprays to prevent respiratory tract infections: a qualitative study of online consumer reviews and primary care patient interviews. BMJ Open. 2022 Jun 30;12(6):e059661. doi: 10.1136/bmjopen-2021-059661. PMID 35772824
- [Background] Slapak I, Skoupa J, Strnad P, Hornik P. Efficacy of isotonic nasal wash (seawater) in the treatment and prevention of rhinitis in children. Arch Otolaryngol Head Neck Surg. 2008 Jan;134(1):67-74. doi: 10.1001/archoto.2007.19. PMID 18209140
- [Background] Tano L, Tano K. A daily nasal spray with saline prevents symptoms of rhinitis. Acta Otolaryngol. 2004 Nov;124(9):1059-62. doi: 10.1080/00016480410017657. PMID 15513550
- [Background] Jaume F, Valls-Mateus M, Mullol J. Common Cold and Acute Rhinosinusitis: Up-to-Date Management in 2020. Curr Allergy Asthma Rep. 2020 Jun 3;20(7):28. doi: 10.1007/s11882-020-00917-5. PMID 32495003